CLINICAL TRIAL: NCT01827631
Title: Single and Repeat Dose Pharmacokinetic Study of GSK1605786 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116416
Record Dates: First submitted 2013-04-05; First posted 2013-04-09 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Crohn's Disease
Keywords: healthy; GSK1605786; CCR9 receptor antagonist; Chinese subjects; pharmacokinetics
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1605786 500 mg once daily (Experimental): GSK1605786 500 mg is given once daily in the morning
  Interventions: Drug: GSK1605786 capsule
- GSK1605786 500 mg twice daily (Experimental): GSK1605786 500 mg is given twice daily in the morning and in the evening
  Interventions: Drug: GSK1605786 capsule

INTERVENTIONS:
Drug: GSK1605786 capsule — Swedish Orange, size 0, hard gelatine capsules

SUMMARY:
This is an open-label, parallel group, single and repeat dose pharmacokinetic (PK) study in healthy male and female subjects. This study will confirm the PK and safety profile in Chinese subjects. GSK1605786 is currently in clinical development for the treatment of Crohn's disease. Subjects will receive one of two GSK1605786 doses (500 mg once daily or 500mg twice daily) within 30 minutes after a meal. The study will consist of single and repeat dose sessions, with pre-dose and serial PK samples taken up to 72-h post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG
* Male or female between 18 and 45 years of age
* Body weight 50 kg (110lbs) for men and women, and body mass index (BMI) within the range 19 24 kg/m2

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary
* A positive test for HIV antibody at screening
* Known coeliac disease and positive serologic testing for anti-tTG antibodies
* A positive pre-study drug/alcohol screen
* Lactating females

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05-27 (Actual); Primary Completion 2013-06-14 (Actual); Study Completion 2013-06-25 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 72 hour post dose
  maximum concentration after single dose and repeat dose
AUC(0-τ) | up to 24 hour post last dose
  area under the concentration time curve during steady state

SECONDARY OUTCOMES:
adverse events (AEs) | up to 21 days, from the first dose until the follow-up visit
  AEs occur during the study
vital signs | before each morning dose on Day 1 and 8-14, and on Day 17 prior to leaving the clinic
  blood pressure, pulse rate, respiratory rate and temperature
lab assessment | Day 17 prior to leaving the clinic
  Hematology/Clinical Chemistry/Urinalysis test

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116416 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116416?search=study&search_terms=116416#rs
- Available data/document: Individual Participant Data Set: 116416 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116416 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116416 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116416 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116416 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116416 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116416 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register